CLINICAL TRIAL: NCT07385365
Title: A Phase Ⅲ Randomized Clinical Study and Real World Study of Postoperative Regional Nodal Radiotherapy in Intermediate-risk Breast Cancer
Brief Title: A Study of Postoperative Regional Nodal Radiotherapy in Intermediate-risk Breast Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shulian Wang,MD, M.D., Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC4876
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; intermediate-risk
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regional nodal irradiation (Experimental): woman with intermediate-risk Breast Cancer involve postoperative conventional fraction/moderate hypofraction/ultrahypofraction radiotherapy to the whole breast/Chest Wall and nodal region
  Interventions: Radiation: Regional nodal Radiotherapy
- Non-Regional nodal irradiation (Active Comparator): woman with intermediate-risk Breast Cancer receive conventional fraction/moderate hypofraction/ultrahypofraction radiotherapy to the whole breast/Chest Wall after breast-conserving surgery or receive no radiotherapy modified radical operation.
  Interventions: Radiation: Non-Regional nodal Radiotherapy

INTERVENTIONS:
Radiation: Regional nodal Radiotherapy — postoperative conventional fraction/moderate hypofraction/ultrahypofraction radiotherapy to the whole breast/Chest Wall and nodal region
  Arms: Regional nodal irradiation
Radiation: Non-Regional nodal Radiotherapy — conventional fraction/moderate hypofraction/ultrahypofraction radiotherapy to the whole breast/Chest Wall after breast-conserving surgery or receive no radiotherapy modified radical operation.
  Arms: Non-Regional nodal irradiation

SUMMARY:
The research hypothesis is that the tumor-free survival rate of intermediate-risk breast cancer patients exempted from RNI is not inferior to that of those receiving RNI. Patients with intermediate-risk breast cancer have a relatively low local-regional recurrence rate whether they undergo RNI or not.Patients were randomly assigned to the RNI group and the non-RNI group.After radiotherapy,the patients are followed the efficacy and toxicities of radiotherapy are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 or above
* Undergo breast-conserving surgery or total mastectomy and axillary lymph node dissection or sentinel lymph node biopsy
* The surgical margin was negative
* Tumor stage:Patients who receive direct surgery : pT1-2N1M0, with at least one lymph node having macrometastasis and a tumor risk score of 0-2.For those who underwent surgery after neoadjuvant chemotherapy: cT1-2N1-2M0→ypT0-2N0M0 (cN+ with pathological confirmation), neoadjuvant Chemotherapy for ≥6 cycles.

Exclusion Criteria:

* distant metastasis
* metastasis of ipsilateral internal mammary, supraclavicular or subclavian lymph nodes
* Had received chest radiotherapy in the past
* Bilateral breast cancer
* Pregnancy or lactation period
* Other malignant tumors in the past or at the same time, and the tumor-free survival time is less than 5 years (excluding non-malignant melanoma skin cancer, papillary thyroid carcinoma/follicular carcinoma, cervical carcinoma in situ)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 3142 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2032-12-31 (Estimated); Study Completion 2042-12-31 (Estimated)

PRIMARY OUTCOMES:
tumor-free survival rate | 5 year

SECONDARY OUTCOMES:
localregional recurrence | 5 year
overall survival | 5 year
acute toxicity | 6 months
late complication | 5 year

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital,Chinese Academy od Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No